CLINICAL TRIAL: NCT04666818
Title: Efficacy of Flash Glucose Monitoring in Pregnant Women With Poorly Controlled Pregestational Diabetes (FlashMom): A Randomized Pilot Study
Brief Title: Efficacy of FGM in Pregestational Diabetes
Acronym: FlashMom
Status: Completed | Type: Observational
Sponsor: University of Catania (Other)
Responsible Party: Principal Investigator, Laura Sciacca, Associate Professor, University of Catania
Other Study IDs: FlashMomStudy
Record Dates: First submitted 2020-11-26; First posted 2020-12-14 (Actual); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Diabetes Mellitus in Pregnancy
Keywords: Flash glucose monitoring; Pregestational diabetes; Glucose control; HbA1c; Glycemic variability; Adverse pregnancy outcomes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Self Monitoring Blood Glucose (SMBG): Women used self-monitoring of blood glucose= Control group (CG)
- Flash Glucose Monitoring (FGM): Women used flash glucose monitoring= FGM group (FG)
  Interventions: Device: Use of Flash Glucose Monitoring

INTERVENTIONS:
Device: Use of Flash Glucose Monitoring — Participants in the intervention group were advised to monitor glucose levels by means of flash glucose system.
  Groups: Flash Glucose Monitoring (FGM)

SUMMARY:
Diabetes is the most common metabolic disease complicating pregnancy, and the number of women in childbearing age facing this problem is rising worldwide. The clinical and social significance of pre-gestational diabetes has become an important issue in the area of public health because this disease can cause maternal complications and influence the development of the offspring during the pregnancy and later in life. Pregnancy in women with pregestational diabetes is indeed associated with adverse perinatal outcomes including large-for gestational- age infants (ranging from 48.8 to 62.5%), preterm delivery, and other perinatal complications. Large-for-gestational-age infants to mothers with diabetes are at increased risk for birth trauma, transient tachypnea, and neonatal hypoglycemia. For all these reasons, the medical costs and social burdens caused by this disease are problematic. The mainstay of managing diabetes during pregnancy is glucose monitoring. Conventionally, glucose monitoring is by self-monitoring of blood glucose (SMBG) involving multiple pricks to the patients. The limitations of these pricks include pain and a point-in-time assessment without evaluation of the complete glycemic profile before making therapeutic adjustments.

Introduction of continuous glucose monitoring (CGM) by measuring interstitial fluid glucose has overcome the deficits in SMBG by providing an overview of the glycemic profiles in patients. In most recent years another promising tool became available: the Flash Glucose Monitoring (FGM) system. Unlike traditional sensor systems, its wired enzyme sensor is calibrated in the factory and therefore requires no user calibrations (fingerstick blood glucose measurements) during the 14 days of wear. Recent studies demonstrated that FGM is effective in reducing glucose fluctuations and preventing hypoglycemic events in Type 1 and Type 2 diabetic patients. No evidence is to date available on the efficacy of FGM on the reduction of the perinatal adverse outcomes during pregnancy in women with pre-gestational diabetes.

The investigators propose to randomize a group of women with poorly controlled pregestational diabetes to receive SMBG (standard antenatal care) or FGM plus SMBG during pregnancy.

DETAILED DESCRIPTION:
Specific Aims Aim 1: To compare the glycemic control and glucose variability during pregnancy and at first postpartum visit in the two randomized groups. This was accomplished by the evaluation of the mean glycated hemoglobin (HbA1c) levels and of several glucose variability indices during gestation and 1 month after delivery. Hypothesis: the real-time information provided by the FGM system improves glucose control and glycemic excursions during pregnancy and after delivery.

Aim 2: To compare the maternal and neonatal adverse outcomes in the two randomized groups at the time of delivery. This was accomplished by the evaluation of the rate of all the most important maternal and fetal-neonatal adverse outcomes (e.g. cesarean section, macrosomia, neonatal hypoglycemia) at the end of gestation. Hypothesis: the use of FGM reduces the rates of those adverse pregnancy outcomes related to maternal hyperglycemia.

Significance and Background Pre-gestational diabetes is still associated with adverse perinatal outcomes largely attributed to maternal hyperglycemia. The risk of adverse outcomes increases with HbA1c higher than 6-6.5% during gestation. Conversely, mean HbA1c levels <6% during the second and third trimester are associated with better outcomes and with the lowest risk of large-forgestational-age infants. Unfortunately, this goal is often difficult to achieve during pregnancy considering that approximately 60% of all pre-gestational diabetic women are poorly controlled at the time of conception and that maternal hypoglycemia should be avoided. Fasting and post-prandial SMBG are recommended in pre-gestational diabetic women to achieve glycemic control during gestation. Additional useful information on direction, frequency and duration of glycemic oscillations could be provided by the CGM. This system, in fact, allows the patients to prevent hypoglycemia and to reduce glucose oscillations measuring interstitial glucose levels continuously. Despite initial controversial results on the efficacy of the CGM technology during pregnancy, a recently published trial demonstrated that Real-Time use of CGM is associated with improved neonatal outcomes (which are likely to be attributed to reduced exposure to maternal hyperglycemia).

Unfortunately the existing CGM devices still need to be frequently calibrated, using a minimum of 2-5 daily monitored capillary blood glucose. The recent introduction of FGM using the factory-calibrated meter has emerged as a novel method to study glycemic patterns. FGM does not require finger prick calibration. The data are extrapolated using the inbuilt software to summarize the glycemic variability over 2 weeks. The glucose profile obtained using this system is called Ambulatory Glucose Profile (AGP). The usefulness of AGP has been studied in adults and pediatric patients affected by diabetes.

Nevertheless, to date there are no studies looking into the efficacy of this tool in women affected by pre-gestational (Type 1 and Type 2) diabetes during pregnancy. The investigators aim to evaluate the effectiveness of antenatal FGM on maternal glycemic control and pregnancy related morbidity in the offspring of mothers with poorly controlled Type 1 and Type 2 diabetes at the time of conception (peri-conception HbA1c ≥6.5%).

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with pregestational diabetes
* HbA1c >6.5%

Exclusion Criteria

* Gestational Diabetes
* HbA1c <6.5%

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators carried out a multicenter randomized pilot trial by prospectively recruiting poorly controlled (peri-conception HbA1c >6.5%) pregestational T1D or T2D outpatients in 5 Italian Diabetes Medical Centers. Enrolling Centers were selected on the basis of the experience in following women with pregestational diabetes and on the presence of the neonatal intensive care unit.
  Randomization was electronically generated at the first pregnancy visit according to a predefined randomization sequence. Women were assigned to either the control group (CG, using the standard SMBG at least 6 times daily) or Flash group (FG, using the FGM system continuously throughout gestation) in a 1:1 ratio.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-11-26 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2020-11-26 (Actual)

PRIMARY OUTCOMES:
Glycosylated Hemoglobin (HbA1c) concentration in blood samples | 38 weeks
  To compare the efficacy of FGM on HbA1c reduction during pregnancy
coefficient of variation (CV): Adimensional coefficient calculated as the Standard Deviation divided by the mean of all glucose values expressed | 33 weeks
  To compare the efficacy of FGM on glucose CV reduction during pregnancy
Mean amplitude of glycemic excursions (MAGE)= Adimensional coefficient calculated mean amplitude of glycemic excursions | 33 weeks
  o compare the efficacy of FGM on MAGE reduction during pregnancy
Continuous overlapping net glycemic action (CONGA)= Adimensional coefficient calculated at 1 hour time interval | 33 weeks
  To compare the efficacy of FGM on CONGA reduction during pregnancy
MODD= Adimensional coefficient calculated as mean of the daily serum glucose difference. | 33 weeks
  To compare the efficacy of FGM on MODD reduction during pregnancy

SECONDARY OUTCOMES:
Macrosomia: Birth weight above 4000 grams regardless gestational age | At birth
  Rate of macrosomic newborn
Large for Gestational Age (LGA)= weight at birth above the 90th percentile for gestational age | At birth
  Rate of LGA newborn
Neonatal Hypoglycemia= plasma glucose level of less than 36 mg/dl | At birth
  Rate of neonatal hypoglycemia
Premature delivery: <37 weeks of gestation | At birth
  Rate of premature delivery
Cesarean section | At delivery
  Rate of Cesarean section

CONTACTS AND LOCATIONS:
Overall Officials: Laura Laura, MD, PhD, Principal Investigator — University of Catania
Locations (1):
- University of Catania, Endocrinology Section, Garibaldi-Nesima Hospital, Catania, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tumminia A, Milluzzo A, Festa C, Fresa R, Pintaudi B, Scavini M, Vitacolonna E, Napoli A, Sciacca L. Efficacy of flash glucose monitoring in pregnant women with poorly controlled pregestational diabetes (FlashMom): A randomized pilot study. Nutr Metab Cardiovasc Dis. 2021 Jun 7;31(6):1851-1859. doi: 10.1016/j.numecd.2021.03.013. Epub 2021 Mar 24. PMID 33975741